CLINICAL TRIAL: NCT07066787
Title: Somatic Symptoms and Depression in Undergraduate Physiotherapy Students: A Community-Based Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, Researcher, Cairo University
Other Study IDs: EGPHYSIO-SC-001
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Somatic Disorders; Psychologic; Public Health
MeSH Terms: interventions — Diploidy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: psychological group — fill the psychological section
Diagnostic Test: somatic — fill the somatic section

SUMMARY:
This cross-sectional, community-based study aimed to investigate the association between depression and somatic symptoms among physical therapy students in Egypt. Using validated tools-the PHQ-9 for depression and PHQ-15 for somatic symptoms-data were collected from undergraduate students through an online questionnaire distributed via social media. The study included students aged 19 to 24 from various Egyptian governorates. Results revealed a notable correlation between depressive symptoms and the severity of physical complaints, highlighting the need for increased mental health support and early screening strategies within physical therapy education programs.

DETAILED DESCRIPTION:
This study is a cross-sectional, community-based investigation designed to explore the relationship between depressive symptoms and somatic complaints among undergraduate physical therapy students in Egypt. Given the increasing academic and psychological pressures faced by health sciences students, particularly those in physically and mentally demanding fields such as physiotherapy, understanding how mental health issues manifest physically is essential for early identification and intervention.

The study was conducted over one week in February 2025, shortly after the start of the academic semester. Participants were recruited through a self-administered online questionnaire shared via social media platforms. The inclusion criteria focused on physical therapy students aged 19 to 24 years, currently enrolled in Egyptian universities. Exclusion criteria included prior psychiatric diagnosis, chronic physical illness, and incomplete responses.

Data collection tools included the Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms and the Patient Health Questionnaire-15 (PHQ-15) to assess the severity and frequency of somatic symptoms. Demographic data and potential influencing factors such as relationship status and plans for part-time work were also recorded.

Ethical approval was obtained from the EG PHYSIO Scientific Committee (Approval Number: EGPHYSIO-SC-001), and the study was registered on ClinicalTrials.gov (Registration ID: NCT06820814). Statistical analysis was performed using SPSS Version 22, with correlation tests used to examine the association between depression scores and somatic symptom severity. Findings from this study aim to inform future strategies for mental health screening, academic support services, and targeted interventions for physiotherapy students in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Medical students currently enrolled in Egyptian universities (public or private).
* Aged between 19 and 24 years.
* Able to read and understand Arabic or English.
* Provided informed consent to participate in the study.
* Completed all sections of the online questionnaire.

Exclusion Criteria:

* Students previously diagnosed with a major psychiatric disorder (e.g., bipolar disorder, schizophrenia).
* Students with chronic physical illnesses that may independently cause somatic symptoms (e.g., fibromyalgia, inflammatory bowel disease).
* Incomplete or duplicate responses to the online questionnaire. Participants who declined to provide informed consent.

Ages: 19 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: The study population consisted of undergraduate physical therapy students currently enrolled in Egyptian universities, both public and private. Participants were between 19 and 24 years of age and represented various academic levels and geographic regions across Egypt. All participants were required to have the ability to read and understand Arabic or English, and to provide informed consent prior to participation. The population was selected to reflect the typical demographic and academic profile of physical therapy students in Egypt, aiming to provide insights into the mental and physical health challenges they face during their education.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 7 days
  assess depressive symptoms
Patient Health Questionnaire-15 (PHQ-15) | 7 days
  assess the severity and frequency of somatic symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Eg Physio, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No